CLINICAL TRIAL: NCT03828838
Title: Pilot Study: Lutetium-177-PSMA-617 in Low Volume Metastatic Prostate Cancer
Brief Title: Lutetium-177-PSMA-617 in Low Volume Metastatic Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL62774.09L.r7
Record Dates: First submitted 2019-01-09; First posted 2019-02-04 (Actual); Last update posted 2019-11-14 (Actual); Status verified 2019-01

CONDITIONS: Prostate Neoplasm
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Pluvicto

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Lu-177 PSMA-617 (Experimental): Two cycles with 3 and 3-6 GBq Lu-177 PSMA-617 (including 3D-dosimetry)
  Interventions: Drug: Lu-177 PSMA-617

INTERVENTIONS:
Drug: Lu-177 PSMA-617 — Two cycles of Lu-177 PSMA (3GBq and 3-6 GBq)
  Other Names: Lutetium-177 Prostate Specific Membrane Antigen

SUMMARY:
Radioligand therapy (RLT) using Lu-177 labelled PSMA is a promising new therapeutic approach to treat metastatic prostate cancer. This tumor-specific treatment is directed against prostate-specific membrane antigen (PSMA), which is overexpressed in prostate cancer cells. In the last few years, several lutetium-177 (177Lu, β emitter) labeled PSMA ligands have been developed and are currently applied to treat metastatic castrate resistant prostate cancer (mCRPC) patients. However, there are no prospective studies published so far using this treatment approach in hormone sensitive setting. In this pilot study patients with hormone sensitive prostate cancer who did not undergo hormonal treatment will be treated with Lu-177 PSMA-617.

DETAILED DESCRIPTION:
Radioligand therapy (RLT) is a promising new therapeutic approach to treat metastatic prostate cancer. This tumor-specific treatment is directed against prostate-specific membrane antigen (PSMA), which is overexpressed in prostate cancer cells. In the last few years, several lutetium-177 (177Lu, β emitter) labeled PSMA ligands have been developed and are currently applied in nuclear medicine departments world-wide to treat metastatic castrate resistant prostate cancer (mCRPC) patients.

A large retrospective study reported an overall biochemical response rate of 45% following multiple 177Lu-PSMA RLT cycles in mCRPC patients, while 40% of patients already responded after a single cycle. RLT with PSMA ligand PSMA-617 was generally well tolerated and 12% of the patients suffered grade 3 to 4 hematological toxicity. In addition, mild and often transient xerostomia occurred in 8%. These results were confirmed in a smaller scale prospective study published recently.

Although these results are very promising, it is noteworthy that all currently Lu-177-PSMA-617 RLT only has been evaluated in end stage prostate cancer patients to date. In theory, RLT could be more effective in low volume disease because of the very high tumor uptake of radioligands in small lesions. There are no published data so far evaluating the therapeutic effect of Lu-177-PSMA-617 RLT in an earlier stage of the disease. Because of the difference in tumor load between mCRPC patients and patients with low volume metastatic disease, dosimetry and toxicity in these patients need evaluation. Here a clinical trial to investigate the efficacy of Lu-177-PSMA-617 RLT in patients with low volume metastatic prostate cancer, prior to the hormone insensitive state is proposed.

Objective: The aim of this study is to evaluate the dosimetry and toxicity of Lu-177-PSMA-617 RLT, in patients with low volume, hormone sensitive metastatic prostate cancer under treatment condition. Ultimately, the goal of this study is to stabilize previously progressive disease in these patients and to improve the quality of life by postponing the need for androgen deprivation therapy (ADT).

ELIGIBILITY:
Inclusion Criteria:

* Histological proven adenocarcinoma of the prostate
* Prior local therapy for prostate cancer
* Biochemical recurrence or clinical progression after local therapy (PSA > 0.2 µg/l),
* PSA-DT < 6 months
* Gallium-68 (68Ga)-PSMA-PET-CT positive metastases in bones and/or lymph nodes (N1/M1ab): ≥1, maximally 10 metastases (at least 1 lesion with a lesion size of ≥1 cm to enable adequate dosimetry studies)
* Local treatment for oligo-metastases with radiotherapy or surgery appears to be no option anymore (due to prior treatment or the location of the metastatic lesions)
* No prior hormonal therapy or chemotherapy; testosteron > 1.7 nmol/l. Exception: local prostate cancer treated with local radiotherapy plus adjuvant ADT; these patients need to be stopped with ADT at least 3 months
* No visceral metastases
* Laboratory values:

  * White blood cells > 3.5 x 109/l
  * Platelet count > 150 x 109/l
  * Hemoglobin > 6 mmol/l
  * Alanine transaminase, aspartate aminotransferase < 3 x upper limit of normal
  * Modification of Diet in Renal Disease Study glomerular filtration rate ≥ 60 ml/min
* Signed informed consent

Exclusion Criteria:

* No detectable lesions on the Ga-68 PSMA PET/CT with an uptake level below the liver uptake.
* A known subtype other than prostate adenocarcinoma
* Any medical condition present that in the opinion of the investigator will affect patients' clinical status when participating in this trial.
* Prior hip replacement surgery potentially influencing performance of PSMA PET/CT and nano Magnet Resonance Tomography (nMRI)
* Contra-indication for MRI imaging (claustrophobia, implanted electric and electronic devices (heart pacemakers, insulin pumps, implanted hearing aids, neurostimulators), intracranial metal clips, metallic bodies in the eye)
* Contra-indication for Buscopan (allergy to hyoscine or any other ingredients of this medication, allergy to to other atropines (e.g. atropine, scopolamine), myasthenia gravis, enlarged colon, glaucoma or obstructive prostatic hypertrophy)
* Additional contra-indications for the intravenous injection form of Buscopan (taking blood thinning medication (e.g. warfarin, heparin), narrowing of the gastrointestinal tract, fast heartbeat, angina or heart failure)
* Contra-indication to glucagon (pheochromocytoma)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-07-01 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Doses delivered to the tumors | For cycle 1 (duration of one cycle is 56 days)
  Calculation of the doses given in Gray per gigabequerel (Gy/GBq) delivered to the tumors
Doses delivered to the tumors | For cycle 2 (duration of one cycle is 56 days)
  Calculation of the doses given in Gray per gigabequerel (Gy/GBq) delivered to the tumors
Doses delivered to organs at risk | For cycle 1 (duration of one cycle is 56 days)
  Calculation of the doses given in Gray per gigabequerel (Gy/GBq) delivered to all organs at risk
Doses delivered to organs at risk | For cycle 2 (duration of one cycle is 56 days)
  Calculation of the doses given in Gray per gigabequerel (Gy/GBq) delivered to all organs at risk

SECONDARY OUTCOMES:
PSA progression free survival | Baseline, at the end of cycle 1 and 2 (each cycle is 28 days) and 3 and 6 months after last cycle
  PSA progression free survival, defined as the time from baseline to PSA progression, assessed using PCWG3 criteria on blood test results.
Uptake on prostate specific membrane antigen (PSMA) positron emission tomography (PET) | Baseline, at the end of cycle 1 and 2 (each cycle is 28 days) and 3 and 6 months after last cycle
  Comparing the changes on baseline PSMA PET and after each cycle (defined according to EORTC PET response criteria)
Radiographic progression free survival | Baseline, at the end of cycle 1 and 2 (each cycle is 28 days) and 3 and 6 months after last cycle
  Radiographic progression free survival - defined as the time from baseline to radiographic progression (assessed using Prostate Cancer Working Group 3 (PCWG3) criteria for bone lesions and RECIST 1.1 for soft tissue lesions)
Health-related quality of life | Baseline, at the end of cycle 1 and 2 (each cycle is 28 days) and 3 and 6 months after last cycle
  Health-related quality of life, assessed using a composite of the European Organisation of Research and Treatment of Cancer (EORTC) core quality of life questionnaire (QLQ C-30)

CONTACTS AND LOCATIONS:
Overall Officials: James Nagarajah, Prof., Principal Investigator — Radboudumc, Nijmegen, Nederland
Locations (1):
- Radiology and Nuclear Medicine, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peters SMB, Mink MCT, Prive BM, de Bakker M, de Lange F, Muselaers CHJ, Mehra N, Witjes JA, Gotthardt M, Nagarajah J, Konijnenberg MW. Optimization of the radiation dosimetry protocol in Lutetium-177-PSMA therapy: toward clinical implementation. EJNMMI Res. 2023 Jan 24;13(1):6. doi: 10.1186/s13550-023-00952-z. PMID 36692682
- [Derived] Prive BM, Peters SMB, Muselaers CHJ, van Oort IM, Janssen MJR, Sedelaar JPM, Konijnenberg MW, Zamecnik P, Uijen MJM, Schilham MGM, Eek A, Scheenen TWJ, Verzijlbergen JF, Gerritsen WR, Mehra N, Kerkmeijer LGW, Smeenk RJ, Somford DM, van Basten JA, Heskamp S, Barentsz JO, Gotthardt M, Witjes JA, Nagarajah J. Lutetium-177-PSMA-617 in Low-Volume Hormone-Sensitive Metastatic Prostate Cancer: A Prospective Pilot Study. Clin Cancer Res. 2021 Jul 1;27(13):3595-3601. doi: 10.1158/1078-0432.CCR-20-4298. Epub 2021 Apr 21. PMID 33883176